CLINICAL TRIAL: NCT00196352
Title: A Prospective, Multiple Site Study to Evaluate the Safety of an Extended Cycle Combination Oral Contraceptive, Seasonique, Which Utilizes Ethinyl Estradiol During the Pill-free Interval.
Brief Title: A Multicenter Study to Evaluate the Safety of Seasonique, an Oral Contraceptive.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PSE-304
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Contraception
Keywords: oral contraceptives; birth control; ethinyl estradiol; pregnancy prevention
MeSH Terms: interventions — Seasonique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Levonorgestrel/EE 0.15/0.03 mg and EE 0.01 mg tablets

INTERVENTIONS:
Drug: Levonorgestrel/EE 0.15/0.03 mg and EE 0.01 mg tablets — 1 tablet daily
  Other Names: Seasonique

SUMMARY:
This study is being conducted to evaluate the safety of ethinyl an extended-regimen oral contraceptive, with ethinyl estradiol supplementation during the usual hormone-free week, for up to an additional three consecutive years.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the safety of an extended-regimen oral contraceptive, with ethinyl estradiol supplementation during the usual hormone-free week, for up to an additional three consecutive years. This is an extension of the Seasonique Phase 3 clinical trial to evaluate long-term safety. Only patients enrolled in the earlier trial are eligible for participation.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the earlier Phase 3 Seasonique clinical trial

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2003-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Patient and Investigator reports of adverse events | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (11):
- United States (11):
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Washington D.C., District of Columbia
  - Duramed Investigational Site, Lincoln, Nebraska
  - Duramed Investigational Site, Rochester, New York
  - Duramed Investigational Site, Charlotte, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Nashville, Tennessee
  - Duramed Investigational Site, Arlington, Virginia
  - Duramed Investigational Site, Norfolk, Virginia